CLINICAL TRIAL: NCT01077791
Title: Cognitive Remediation of the Ability to Infer Intention of Others in Schizophrenic Patients - A Controlled, Randomized Trial (Phase IIb)
Brief Title: A Study of a Remediation Program of Social Cognition in Schizophrenia
Acronym: REMEDCOG
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: no reponse of the of the treatment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P070112; 2007-A00916-47 (Registry Identifier: idrcb)
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2010-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; social cognition; theory of mind; cognitive therapy; therapeutic trial; magnetoencephalography (MEG)
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- original cognitive therapy (Experimental)
  Interventions: Behavioral: original cognitive therapy
- no intervention (No Intervention)

INTERVENTIONS:
Behavioral: original cognitive therapy — 12 weekly sequences of an original cognitive therapy based on videos involving the learning of a better use of contextual information to infer others' intention. Group of 5 patients trained by 2 therapeutics. Comparison with a non-cognitive psychoeducational training (same organisational design).
  Arms: original cognitive therapy

SUMMARY:
Theory of mind (ability to infer others' intention, emotion, etc) is known to be altered in patients with schizophrenia and its deficit to be correlated with their decreased social proficiency. We designed a novel cognitive therapy, that makes use of videos, aimed at learning a better use of contextual information to infer others' intentions. The aim of this study is to demonstrate, in schizophrenic patients, a quantitative improvement of their ability to infer intention of others induced by this novel training program. A secondary aim is to measure the cerebral correlates (MEG, PeV) of this social cognitive function and of its anticipated improvement.

DETAILED DESCRIPTION:
Scientific justification : Improvement by training has been demonstrated in Schizophrenic patients for various cognitive functions and skills, though not yet for the social cognition ability specifically dedicated to infer others' intention when not explicit.

Main hypothesis : Abilities to infer other's intention can improve in schizophrenic patients following specific practice.

Primary aim : To demonstrate this improvement, as quantified by improvement of V-SIR scores (V-LIS scores in French literature).

Procedure : Ten weekly sessions of a novel cognitive therapy that makes use of videos aimed at learning a better use of contextual information to infer others' intentions. Group of 5 patients trained by 2 therapists. Comparison with a non-cognitive psycho-educational training (same organisational design).

Study design : Controlled randomized simple blind study (equivalent to a Phase IIb therapeutic trial). Matched pair design. 40 patients (20 per arm).

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia following DSM IV;
* Age 18-57;
* Stability of the clinical state;
* Ability to learn;
* Deficit in intention reading as measure with the V-SIR (V-LIS in French) test (score >13);
* informed consent to participate to the study.

Exclusion Criteria:

* Any other organic or neuropsychiatric disease

Ages: 18 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate a measurable improvement of Theory of Mind based ability in schizophrenic patients induced by a novel cognitive therapy, as quantified by improvement of V-SIR scores (V-LIS scores in French literature). | 6 MONTHS

SECONDARY OUTCOMES:
To measure the extension of improvement to other cognitive functions - specific or non specific - and/or to every day life aptitudes | 6 MONTHS
To evaluate correlations with functional measurements (e.g., magneto-encephalography, cognitive evoked potentials) [transversal study; longitudinal study]. | 6 MONTHS

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Bourdet, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre hospitalier de Versailles. Service de Psychiatrie., Le Chesnay, France